CLINICAL TRIAL: NCT06713278
Title: Association Between Tension-Type Headache and Masseter Muscle Thickness in Women with Fibromyalgia
Brief Title: Tension-Type Headache and Masseter Thickness in Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Handan Elif Nur BAYRAKTAR, Specialist, Erol Olcok Corum Training and Research Hospital
Other Study IDs: CORUM-PMR-DRHENY-01
Record Dates: First submitted 2024-11-24; First posted 2024-12-03 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Fibromyalgia
Keywords: tension type headache; masseter muscle
MeSH Terms: conditions — Fibromyalgia; Tension-Type Headache | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- fibromyalgia with tension type headache: fibromyalgia with tension type headache
  Interventions: Other: masseter muscle thickness measurement; Other: scales
- fibromyalgia without tension type headache: fibromyalgia without tension type headache
  Interventions: Other: masseter muscle thickness measurement; Other: scales
- control group: control group
  Interventions: Other: masseter muscle thickness measurement; Other: scales

INTERVENTIONS:
Other: masseter muscle thickness measurement — masseter muscle thickness measurement with ultrasonography
Other: scales — headache impact scale (HIT-6) Short SF-36 fibromyalgia total score widespread pain index symptom severity scale fibromyalgia impact questionnaire (FIQ)

SUMMARY:
This study aims to investigate the relationship between tension-type headaches and masseter muscle thickness in women with fibromyalgia syndrome (FMS) and to explore the potential for new therapeutic approaches in the treatment of both headaches and FMS. Additionally, the study seeks to evaluate the impact of headaches on the quality of life in individuals with FMS.

Does tension-type headache associate with increased masseter muscle thickness in women with fibromyalgia syndrome (FMS)? Does tension-type headache negatively impact the quality of life in women with FMS?

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is a chronic condition characterized by widespread musculoskeletal pain, fatigue, cognitive dysfunction, and tenderness, affecting approximately 5% of the global population, predominantly women. Central sensitization plays a key role in its pathophysiology. Tension-type headaches, the most common in FMS (59.01%), are associated with pericranial muscle sensitivity, anxiety, and reduced quality of life. Increased masseter muscle activity has been observed in tension-type headaches, but its relationship with FMS remains unexplored.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-65 years.
* Diagnosed with fibromyalgia syndrome (FMS) according to the 2016 American College of Rheumatology (ACR) diagnostic criteria.
* At least one year since the FMS diagnosis.
* Chronic tension-type headache lasting for at least six months.
* Diagnosed with tension-type headache by a neurologist based on the International Classification of Headache Disorders (ICHD-3) criteria.

Exclusion Criteria:

* Patients with neurological or psychiatric disorders.
* Patients using medications related to the central nervous system.
* Those with temporomandibular dysfunction.
* Patients with rheumatologic diseases.
* Individuals undergoing dental treatment or using dental prostheses.
* Those with facial tumors or a history of facial surgery.
* Pregnant women.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: female 18-65 years
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Masseter muscle thickness | 1 day
  Measurement of masseter muscle thickness by ultrasonography

SECONDARY OUTCOMES:
HIT-6 (Headache Impact Test-6) | 1 day
  HIT-6 (Headache Impact Test-6):The HIT-6 (Headache Impact Test-6) consists of 6 questions, each evaluated using a 5-point Likert scale. The scale assigns the following scores: 6 points for "never," 8 points for "rarely," 10 points for "sometimes," 11 points for "very often," and 13 points for "always." The total score ranges from 36 to 78. The severity of the headache's impact is categorized as follows:
  60-78: Severe impact 56-59: Substantial impact 50-55: Moderate impact <49: Little to no impact Higher scores indicate worse outcomes.
FIQ (Fibromyalgia Impact Questionnaire) | 1 day
  FIQ (Fibromyalgia Impact Questionnaire):The Fibromyalgia Impact Questionnaire (FIQ) is a validated and reliable tool in Turkish that measures the impact of fibromyalgia on daily life. It consists of 10 main items covering various aspects of daily life, including physical functionality, ability to perform tasks, sleep quality, emotional well-being, and pain. The total FIQ score is categorized as follows:
  0-38: Mild impact 39-58: Moderate impact 59-100: Severe impact Higher scores indicate worse outcomes.
Fibromyalgia Total Score | 1 day
  The Fibromyalgia Total Score assesses the severity and impact of fibromyalgia symptoms. It is typically calculated as the sum of two components: the Widespread Pain Index (WPI) and the Symptom Severity Scale (SSS).
  Calculation Widespread Pain Index (WPI):Evaluates the number of body regions experiencing pain, ranging from 0 to 19.
  Symptom Severity Scale (SSS):Assesses the severity of fatigue, unrefreshed sleep, and cognitive difficulties, along with the presence of other somatic symptoms, ranging from 0 to 12.
  Total Score:The Fibromyalgia Total Score ranges from 0 to 31. Higher scores indicate more severe symptoms and a greater impact of fibromyalgia. Higher scores indicate worse outcomes.
  This score is used to aid in diagnosing fibromyalgia and evaluating its severity.
Widespread Pain Index (WPI) | 1 day
  The Widespread Pain Score (WPI) is a measure included in the 2016 ACR fibromyalgia diagnostic criteria. It consists of 19 body regions. Participants indicate the areas where they experience pain, receiving 1 point for each marked region. The WPI is scored on a scale of 0 to 19. Higher scores indicate worse outcomes.
Symptom Severity Scale (SSS) | 1 day
  The Symptom Severity Scale (SSS) is a measure included in the 2016 ACR fibromyalgia diagnostic criteria.
  First Section: Evaluates fatigue, waking unrefreshed, and cognitive symptoms, scored as follows:0 (none), 1 (mild), 2 (moderate), 3 (severe).
  Second Section: Assesses the presence of headaches, lower abdominal pain, and depression, scored as:0 (absent), 1 (present).
  The total SSS score ranges from 0 to 12. Higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Çorum Hitit University Erol Olçok Training and Research Hospital, Çorum, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moraska AF, Stenerson L, Butryn N, Krutsch JP, Schmiege SJ, Mann JD. Myofascial trigger point-focused head and neck massage for recurrent tension-type headache: a randomized, placebo-controlled clinical trial. Clin J Pain. 2015 Feb;31(2):159-68. doi: 10.1097/AJP.0000000000000091. PMID 25329141
- [Background] Shields G, Smith JM. Remedial Massage Therapy Interventions Including and Excluding Sternocleidomastoid, Scalene, Temporalis, and Masseter Muscles for Chronic Tension Type Headaches: a Case Series. Int J Ther Massage Bodywork. 2020 Feb 26;13(1):22-31. eCollection 2020 Mar. PMID 32133042
- [Background] Martin-Vera D, Sanchez-Sierra A, Gonzalez-de-la-Flor A, Garcia-Perez-de-Sevilla G, Dominguez-Balmaseda D, Del-Blanco-Muniz JA. Efficacy of a strength-based exercise program in patients with chronic tension type headache: a randomized controlled trial. Front Neurol. 2023 Sep 18;14:1256303. doi: 10.3389/fneur.2023.1256303. eCollection 2023. PMID 37789886
- [Background] de Tommaso M. Prevalence, clinical features and potential therapies for fibromyalgia in primary headaches. Expert Rev Neurother. 2012 Mar;12(3):287-95; quiz 296. doi: 10.1586/ern.11.190. PMID 22364327
- [Background] Lee K, Chon S. Assessments of Muscle Thickness and Tonicity of the Masseter and Sternocleidomastoid Muscles and Maximum Mouth Opening in Patients with Temporomandibular Disorder. Healthcare (Basel). 2021 Nov 26;9(12):1640. doi: 10.3390/healthcare9121640. PMID 34946366
- [Background] Kobayashi R, Haga S, Umehara A, Takakaze M, Akatsuka K, Nakano H. Quantitative and qualitative evaluation of the masseter muscle by ultrasonography and correlation with whole body health status. J Phys Ther Sci. 2024 Mar;36(3):136-141. doi: 10.1589/jpts.36.136. Epub 2024 Mar 1. PMID 38434992
- [Background] Andersen S, Petersen MW, Svendsen AS, Gazerani P. Pressure pain thresholds assessed over temporalis, masseter, and frontalis muscles in healthy individuals, patients with tension-type headache, and those with migraine--a systematic review. Pain. 2015 Aug;156(8):1409-1423. doi: 10.1097/j.pain.0000000000000219. PMID 25955963
- [Background] Alizadeh Savareh B, Ghanjal A, Bashiri A, Motaqi M, Hatef B. The power features of Masseter muscle activity in tension-type and migraine without aura headache during open-close clench cycles. PeerJ. 2017 Jul 25;5:e3556. doi: 10.7717/peerj.3556. eCollection 2017. PMID 28775915
- [Background] May A. Hints on Diagnosing and Treating Headache. Dtsch Arztebl Int. 2018 Apr 27;115(17):299-308. doi: 10.3238/arztebl.2018.0299. PMID 29789115
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Background] Nielsen LA, Henriksson KG. Pathophysiological mechanisms in chronic musculoskeletal pain (fibromyalgia): the role of central and peripheral sensitization and pain disinhibition. Best Pract Res Clin Rheumatol. 2007 Jun;21(3):465-80. doi: 10.1016/j.berh.2007.03.007. PMID 17602994
- [Background] Siracusa R, Paola RD, Cuzzocrea S, Impellizzeri D. Fibromyalgia: Pathogenesis, Mechanisms, Diagnosis and Treatment Options Update. Int J Mol Sci. 2021 Apr 9;22(8):3891. doi: 10.3390/ijms22083891. PMID 33918736